CLINICAL TRIAL: NCT01802827
Title: Ventilator Associated Tracheobronchitis in the First 14 Days in ICU
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Efstratios Manoulakas, Ph, Principal Investigator, University of Thessaly
Other Study IDs: MARKAR236
Record Dates: First submitted 2012-09-24; First posted 2013-03-01 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Airway Colonization; Tracheobronchitis and Pneumonia Associated With Ventilator
Keywords: airway colonization; tracheobronchitis; pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, sputum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- VAT patients: Patients developing Ventilator Associated Tracheobronchitis
- VAP: Patients presenting ventilator associated pneumonia
- No ventilator associated infection: patients who do not present ventilator associated infection during their stay in ICU

SUMMARY:
To investigate the clinical course and risk factors for VAT and the impact of VAT on Intensive Care Unit (ICU) morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* > 48 hours mechanical ventilation

Exclusion Criteria:

* immunodeficiency
* pregnancy
* severe COPD, chronic bronchitis, bronchiectasis
* recent pneumonia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients ventilated > 48hours
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
mortality | mortality at 4 weeks
  we assessed mortality from all causes at 4 weeks

SECONDARY OUTCOMES:
ICU length of stay | expected average length of stay 15 days
mortality at 6 months | 6 months